CLINICAL TRIAL: NCT02637778
Title: Intervention Study - Modulation of Cardiovascular Risk Factors by Personal Nutritional Counselling and Daily Menu Plans
Brief Title: Modulation of Cardiovascular Risk Factors by the Diet
Acronym: MoKaRi-Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Christine Dawczynski,PhD, PhD, University of Jena
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H2_16
Record Dates: First submitted 2015-12-15; First posted 2015-12-22 (Estimated); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Cardiovascular Diseases
Keywords: nutrient profiles; menu plans; n-3 LC-PUFA; SFA; MUFA; PUFA; cardiovascular risk
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cardioprotective diet (Experimental): The study participants receive defined personal nutrition counselling every two weeks and they get daily menu plans (with optimised nutrient profiles) over an entire period of 20 wks (follow-up 20 wks).
  Interventions: Dietary Supplement: Cardioprotective diet
- Cardioprotective diet + 3 g EPA+DHA/d (Experimental): The study participants receive defined personal nutrition counselling every two weeks and they get daily menu plans (with optimised nutrient profiles) over an entire period of 20 wks (follow-up 20 wks).
  Participants will consume additional n-3 LC-PUFA (3 g EPA+DHA/d).
  Interventions: Dietary Supplement: Cardioprotective diet + 3 g EPA + DHA/d

INTERVENTIONS:
Dietary Supplement: Cardioprotective diet — The 'cardioprotective diet' is characterized by (i) adequate energy intake, (ii) intake of carbohydrates, protein, fat according to the guidelines of the German Society of Nutrition (DGE e. V.), (iii) desirable intake of saturated fatty acids (SFA, 7 En%), monounsaturated fatty acids (MUFA, > 10 En%), polyunsaturated fatty acids (PUFA, approx. 10 En%) and in particular n-3 LC-PUFA, (iv) encouraged consumption of vegetables, fruits, cereals, (v) salt and sugar reduction, (vi) avoiding of highly processed, calorie-dense, nutrient-poor food as well as (vii) encouraged physical activity.
  Arms: Cardioprotective diet
Dietary Supplement: Cardioprotective diet + 3 g EPA + DHA/d — The 'cardioprotective diet' is characterized by (i) adequate energy intake, (ii) intake of carbohydrates, protein, fat according to the guidelines of the German Society of Nutrition (DGE e. V.), (iii) desirable intake of saturated fatty acids (SFA, 7 En%), monounsaturated fatty acids (MUFA, > 10 En%), polyunsaturated fatty acids (PUFA, approx. 10 En%) and in particular n-3 LC-PUFA, (iv) encouraged consumption of vegetables, fruits, cereals, (v) salt and sugar reduction, (vi) avoiding of highly processed, calorie-dense, nutrient-poor food as well as (vii) encouraged physical activity.The participants will consume additional n-3 LC-PUFA (3 g EPA+DHA/d)
  Arms: Cardioprotective diet + 3 g EPA+DHA/d

SUMMARY:
The interventional study will evaluate effectiveness and potential of a 'cardioprotective diet' for adults with increased risk for cardiovascular diseases (CVD). The 'cardioprotective diet' is characterized by adequate energy intake, intake of carbohydrates, protein and fat according to the guidelines of the German Society of Nutrition (DGE e. V.), with special focus on fat quality of the foods.

Half of the participants will consume additional n-3 long-chain (LC)-PUFA (3 g eicosapentaenoic acid (EPA) + docosahexaenoic acid (DHA)/d). The study participants receive defined personal nutritional counselling every two weeks and they get daily menu plans (with optimised nutrient profiles) over an entire period of 20 weeks (follow-up 20 weeks).

DETAILED DESCRIPTION:
The interventional study will evaluate effectiveness and potential of a 'cardioprotective diet' for adults with increased risk for cardiovascular diseases (CVD). The 'cardioprotective diet' is characterized by (i) adequate energy intake, (ii) intake of carbohydrates, protein, fat according to the guidelines of the German Society of Nutrition (DGE e. V.), (iii) desirable intake of saturated fatty acids (SFA, 7 En%), monounsaturated fatty acids (MUFA, > 10 En%), polyunsaturated fatty acids (PUFA, approx. 10 En%) and in particular n-3 LC-PUFA, (iv) encouraged consumption of vegetables, fruits, cereals, (v) salt and sugar reduction, (vi) avoiding of highly processed, calorie-dense, nutrient-poor food as well as (vii) encouraged physical activity.

Half of the participants will consume additional n-3 LC-PUFA (3 g EPA+DHA/d). The study participants receive defined personal nutritional counselling every two weeks and they get daily menu plans (with optimised nutrient profiles) over an entire period of 20 weeks (follow-up 20 weeks).

Besides the personal dialogues participants receive information materials providing the dietary recommendations, information to improve nutritional behavior and environment as well as various practical advices. Additionally, a weekly reminder strengthens the approach in addition to each visit at a 2-week interval.

The reflection about the implementation of the advices within day-to-day routine and the resulting challenges are an important part of the concept (feedback).

The identification of variables influencing people's nutritional behavior is attained and offers the possibility to address these variables within the recommendations that will be developed for adults with increased CVD risk as part of our nutriCARD strategy (Competence Cluster for Nutrition and Cardiovascular Health (nutriCARD), Halle-Jena-Leipzig, Germany).

The study will provide data about the association between the defined dietary intake and measurable markers reflecting food intake (nutritional biomarkers) as well as expression of cardiovascular biomarkers.

ELIGIBILITY:
Inclusion Criteria:

- LDL cholesterol ≥ 3 mmol/L

Exclusion Criteria:

* intake of lipid-lowering medications
* gastrointestinal diseases
* familial hypercholesterolemia
* intake of additional dietary supplements (especially fish oil capsules or vitamin E)
* pregnancy, lactation
* patient's request or if patient compliance with the study protocol is doubtful

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
blood lipids | change from baseline at 20 weeks
  total cholesterol, LDL cholesterol, HDL cholesterol, triacylglycerides (TAG) [mmol/L]

SECONDARY OUTCOMES:
fatty acid distribution (blood) | change from baseline at 20 weeks
  Fatty acid distribution in plasma lipids und erythrocyte lipids [% FAME (fatty acid methyl ester)]
insulin (blood) | change from baseline at 20 weeks
  [units/ml]
HbA1c (blood) | change from baseline at 20 weeks
oral glucose tolerance test (blood) | change from baseline at 20 weeks
  blood glucose (timepoints: 0, 60 min, 120 min) after oral challenge (75 g glucose) [mmol/l]
alpha prothrombin time (blood) | change from baseline at 20 weeks
  [sec]
fibrinogen (blood) | change from baseline at 20 weeks
  [g/l]
Nutritional status I (blood) | change from baseline at 20 weeks
  vitamins (A, E), folic acid, iodine [µg/l]
Nutritional status II (blood) | change from baseline at 20 weeks
  vitamin D, vitamin B12 [pg/ml]
Nutritional status III (blood) | change from baseline at 20 weeks
  vitamin B1, B6 [ng/ml]
homocysteine (blood) | change from baseline at 20 weeks
  [µmmol/l]
high sensitive c-reactive protein (blood) | change from baseline at 20 weeks
  [mg/dl]
lipoprotein(a) (blood) | change from baseline at 20 weeks
  [mg/dl]
height | change from baseline at 20 weeks
  [m]
weight | change from baseline at 20 weeks
  [kg]

OTHER OUTCOMES:
apolipoproteins (blood) | change from baseline at 20 weeks
  apolipoprotein A1, apolipoprotein B [g/l]
adiponectin (blood) | change from baseline at 20 weeks
  [mg/l]
leptin, resistin (blood) | change from baseline at 20 weeks
  [µg/l]
creatinine (24h urine) | change from baseline at 20 weeks
  [mmol/24h]
albumin (24h urine) | change from baseline at 20 weeks
  [mg/dl]
Nutritional status IV (24h urine) | change from baseline at 20 weeks
  natrium, magnesium (24h urine) [mmol/24h]
Nutritional status V (24h urine) | change from baseline at 20 weeks
  copper (24h urine) [µg/g creatinine]
Nutritional status VI (24h urine) | change from baseline at 20 weeks
  manganese (24h urine) [µg/l]

CONTACTS AND LOCATIONS:
Overall Officials: Christine Dawczynski, PhD, Principal Investigator — University oj Jena, Department of Nutritional Biochemistry and Physiology; Competence Cluster for Nutrition and Cardiovascular Health (nutriCARD), Halle-Jena-Leipzig, Germany; Stefan Lorkowski, PhD, Principal Investigator — University oj Jena, Department of Nutritional Biochemistry and Physiology; Competence Cluster for Nutrition and Cardiovascular Health (nutriCARD), Halle-Jena-Leipzig, Germany

REFERENCES:
- [Derived] Dawczynski C, Drobner T, Weidauer T, Schlattmann P, Kiehntopf M, Weber D, Grune T, Marz W, Kleber ME, Lorkowski S. Reduction of cardiovascular risk factors by the diet - Evaluation of the MoKaRi concept by a parallel-designed randomized study. Lipids Health Dis. 2025 Mar 8;24(1):88. doi: 10.1186/s12944-025-02500-1. PMID 40057729
- [Derived] Dawczynski C, Cullen PM, Schlattmann P, Lorkowski S. A study protocol of a randomized trial evaluating the effect of using defined menu plans within an intensive personal nutritional counseling program on cardiovascular risk factors: The MoKaRi (modulation of cardiovascular risk factors) trial. Contemp Clin Trials Commun. 2021 Apr 29;22:100761. doi: 10.1016/j.conctc.2021.100761. eCollection 2021 Jun. PMID 33997459
- See also: Study protocoll — https://doi.org/10.1016/j.conctc.2021.100761
- See also: Study results — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7146433/